CLINICAL TRIAL: NCT02743000
Title: Emotion and Reward Processing in Binge Eating
Brief Title: Food and the Brain
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Cara Bohon, PhD, Assistant Professor, Stanford University
Other Study IDs: 35204
Record Dates: First submitted 2016-04-12; First posted 2016-04-19 (Estimated); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Binge Eating
Keywords: fMRI; emotion conflict task; monetary incentive delay
MeSH Terms: conditions — Bulimia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Women ages 18-35: Women ages 18-35 who do and do not engage in binge eating will be included in the study

SUMMARY:
The proposed study will examine the role of reward and emotion in women with and without a history of binge eating. It is important to understand how the brain responds to reward and emotion in binge eating in order to identify different pathways toward binge eating and provide individualized targets for treatment. This is particularly important in light of the fact that for many patients, the current treatments for binge eating are not effective.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Ages 18-35
* with or without current binge eating behaviors

Exclusion Criteria:

* Any contraindication for MRI (orthodontia, vascular stents, metallic ear tubes, metal implants, piercings, etc).
* substance abuse
* traumatic brain injury
* BMI < 18.5
* pregnant women

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women ages 18-35
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2016-01; Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Brain activity during rest | Baseline
  Functional magnetic resonance imaging will be used to measure brain activity at rest and connectivity between brain regions will be examined.
Brain activity during emotion conflict | Baseline
  Functional magnetic resonance imaging will be used to measure brain activity during a task where participants respond to images of faces with emotional expressions overlaid with an emotion word written in text. We will focus on brain response during this task when emotion face vs word are in conflict.
Brain activity during monetary wins and losses | Baseline
  Functional magnetic resonance imaging will be used to measure brain activity during a game where participants can win or lose money if they respond to a shape on the computer screen. Brain response during wins and losses will be examined.

CONTACTS AND LOCATIONS:
Overall Officials: Cara Bohon, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Department of Psychiatry, Stanford, California, United States